CLINICAL TRIAL: NCT00509327
Title: Randomized Clinical Trial of Bisacodyl Versus Placebo on Postoperative Bowel Motility in Elective Colorectal Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2004DR4256
Record Dates: First submitted 2007-07-30; First posted 2007-07-31 (Estimated); Last update posted 2007-07-31 (Estimated); Status verified 2007-04

CONDITIONS: Postoperative Ileus
Keywords: postoperative ileus; colorectal surgery; bisacodyl; laxatives
MeSH Terms: interventions — Bisacodyl

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): bisacodyl 10mg twice daily from one day preoperative to day three postoperative
  Interventions: Drug: bisacodyl
- 2 (Placebo Comparator): 10mg of glucosemonohydricum twice daily from one day preoperative to day three postoperative
  Interventions: Drug: glucosemonohydricum

INTERVENTIONS:
Drug: bisacodyl — 10mg capsule twice daily from one day preoperatively to day three postoperatively
  Arms: 1
Drug: glucosemonohydricum — 10mg of glucosemonohydricum twice daily from one day preoperative to day three postoperative
  Arms: 2

SUMMARY:
Postoperative bowel dysmotility is a frequent condition after colorectal surgery. The influence of colon stimulating laxatives have not been studied. This prospective, randomized, double blind, placebo controlled study assesses the influence of bisacodyl on postoperative bowel motility in patients undergoing elective colorectal surgery. The hypothesis of this trial was that bisacodyl has a beneficial effect on the duration of postoperative ileus.

DETAILED DESCRIPTION:
All adult (>18 years) patients admitted for elective colorectal resection were evaluated for eligibility.

Patients were randomized using a computer programme and received either 10mg of bisacodyl in non-transparent capsules or identical placebo capsules, containing glucosemonohydricum. The capsules were administered twice daily, starting one day before surgery and ending on postoperative day three.Patients and all involved medical personnel were blinded.

Bowel preparation was not routinely used in open surgery, whereas in patients undergoing laparoscopic resection two litres of sodium-sulfate / macrogol solution (Cololyt®, Spirig Pharma AG, Switzerland) was administered. Standard colorectal surgery was performed in all patients. In open surgery a midline incision was used for laparotomy. In laparoscopic resections a four-port technique with removal of the specimen through a small transverse incision in the lower abdomen was used. All patients received perioperative single shot antibiotics, cefuroxime 1.5 g and metronidazole 1g. Nasogastric tube (NGT) was scheduled to be removed at the end of surgery. Postoperative treatment was not changed during the study. All patients received postoperatively a basic analgesia of 500 to 1000 mg oral paracetamol every 6 h; additionally, metamizol was administrated intravenously or orally as needed.

The primary endpoint was the time to recovery of gastrointestinal function, defined as the mean time to the occurrence of the following three events (GI-3): first flatus passed, first defecation and first solid food tolerated. We did not include the presence of bowel movement, as they may be present before recovery of the colon due to small bowel activity24. Secondary endpoints were the incidence of NGT reinsertion, duration of NGS reinsertion, incidence of postoperative vomiting and length of hospital stay. Additionally, consumption of analgesics and pain, cramping and nausea scores (assessed with a visual analogue scale [VAS]) during the first 8 postoperative days were monitored. Other variables recorded were patients' demographics, use of epidural anaesthesia, type and duration of surgery and morbidity.

ELIGIBILITY:
Inclusion Criteria:

* elective colorectal resection
* age >18 years

Exclusion Criteria:

* preoperatively planned stoma formation
* emergency surgery
* pregnancy
* known hypersensitivity for bisacodyl

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2004-11; Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Time to recovery of gastrointestinal function, defined as the mean time to the occurrence of the following three events (GI-3): first flatus passed, first defecation and first solid food tolerated | 10 days

SECONDARY OUTCOMES:
Incidence of NGT reinsertion, duration of NGS reinsertion, incidence of postoperative vomiting and length of hospital stay | 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Urs Zingg, MD, Principal Investigator — department of Surgery, University Hospital Basel, Switzerland; Urs Metzger, Professor, Study Director — Triemli Hospital, Zurich, Switzerland
Locations (1):
- Department of Surgery, Triemli Hospital, Zurich, Switzerland, Zurich, Switzerland